CLINICAL TRIAL: NCT03804554
Title: Nivolumab in the Treatment of Patients With Non-small Cell Lung Cancer: The Australian Experience
Brief Title: A Study of Participants in Australia Who Have Non-small Cell Lung Cancer Being Treated With Nivolumab
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8MH
Record Dates: First submitted 2018-11-12; First posted 2019-01-15 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients taking nivolumab
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study is to capture and describe the patient and disease characteristics and the outcomes of adult patients with previously-treated advanced NSCLC who have been treated with Nivolumab

ELIGIBILITY:
Inclusion Criteria

* Adult male or female (≥18 years of age) patients with NSCLC
* Treated with nivolumab on the Australian PAP
* Initiated Nivolumab between May 2015 and August 2017
* Attending clinician agreeable to provide patient data
* Local institutional ethics requirements satisfied

Exclusion Criteria:

* Insufficient data available

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously-treated advanced NSCLC patients commencing treatment with nivolumab between May 2015 and August 2017 under the Australian Patient Access Program
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) | Approximately 27 months

SECONDARY OUTCOMES:
Best overall response (BOR) | Approximately 27 months
Progression free survival rate (PFSR) | Approximately 27 months
Overall survival rate (OSR) | Approximately 27 months
Incidence of AE's | Approximately 27 months
Incidence of SAE's | Approximately 27 months
Reasons for ceasing treatment | Approximately 27 months
  Any of the following: progressive disease, toxicity, patient wishes/preference, doctor decision, death
Incidence of patients with brain metastases | Approximately 27 months
Incidence of re-treatment | Approximately 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Heidelburg, Victoria, Australia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm